CLINICAL TRIAL: NCT00009646
Title: Trial of Indomethacin Prophylaxis in Preterm Infants (TIPP)
Acronym: TIPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Medical Research Council of Canada (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Barbara Schmidt/ Lead Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0011; U10HD034216 (NIH); U10HD027904 (NIH); U10HD021364 (NIH); U10HD027851 (NIH); U10HD021397 (NIH); U10HD027881 (NIH); U10HD027880 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); MT-13288 (Other Grant/Funding Number: Medical Research Council of Canada); M01RR000997 (NIH); M01RR000070 (NIH)
Record Dates: First submitted 2001-02-01; First posted 2001-02-05 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Very Low Birth Weight; Infant, Premature; Ductus Arteriosus, Patent
Keywords: Chronic lung disease; Indocin; Indomethacin; Infants, very low birth weight; Intraventricular hemorrhage; Necrotizing enterocolitis; Patent ductus arteriosus; Pulmonary hemorrhage
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent; Enterocolitis, Necrotizing | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indomethacin (Experimental): Indocid P.D.A., Merck Frosst, Kirkland, Que., Canada, and Merck, West Point, Pa.
  Interventions: Drug: indomethacin
- Placebo (Placebo Comparator): Saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: indomethacin — Indocid P.D.A., Merck Frosst, Kirkland, Que., Canada, and Merck, West Point, Pa
  Arms: Indomethacin
Drug: Indomethacin — 0.1 mg per kilogram of body weight
  Arms: Indomethacin
Drug: Placebo — 0.1 mg per kilogram of body weight
  Arms: Placebo

SUMMARY:
This trial was to determine whether giving low-dose indomethacin to infants weight 500 to 999 grams (approximately 1 to 2 pounds) at birth improves their survival without cerebral palsy or developmental problems at 18 to 22 months of age.

DETAILED DESCRIPTION:
Prophylactic indomethacin reduces patent ductus arteriosus (PDA) and intraventricular hemorrhage in very low birth weight infants. However, the effects of early indomethacin on long-term neurodevelopment remain uncertain. There is also insufficient evidence to rule out serious adverse effects, such as increases in the risk of necrotizing enterocolitis (NEC) and retinopathy of prematurity (ROP). The aim of this trial was to determine if prophylactic administration of indomethacin improves survival without neurosensory impairments in extremely-low-birth-weight infants. Infants (n=1202) with birthweights 500 to 999 grams were randomized between 2 and 6 hours after birth to receive either intravenous indomethacin (0.1 mg/kg) or equal volumes of normal saline placebo, daily for 3 days. The primary outcomes at a corrected age of 18 months was a composite of death, cerebral palsy, cognitive delay, deafness, or blindness. Secondary long-term outcomes were hydrocephalus necessitating the placement of a shunt, seizure disorder, and microcephaly. Secondary short-term outcomes were patent ductus arteriosus, pulmonary hemorrhage, chronic lung disease, cranial ultrasonographic abnormalities, nectrotizing enterocolitis and retinopathy. Infants were evaluated in follow-up at 18-22 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight 500 to 999 grams;
* Postnatal age greater than 2 hours;

Exclusion Criteria:

* Unable to administer study drug within 6 hours of birth;
* Structural heart disease and/or renal disease;
* Dysmorphic features or congenital abnormalities;
* Tocolytic therapy with indomethacin or other prostaglandin inhibitor within 72 hours prior to delivery;
* Overt clinical bleeding from more than one site;
* Platelet count less than 50 x 109/L;
* Hydrops;
* Not considered viable

Ages: 2 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1202 (Actual)
Dates: Start 1993-11; Primary Completion 1999-03 (Actual); Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Death or Neurodevelopment Impairment | 18-22 Months Corrected Age

SECONDARY OUTCOMES:
Patent ductus arteriosus | 120 Days of Life
Bronchopulmonary Dysplasia (BPD) | 120 Days of Life
  Chronic Lung Disease (CLD)
Necrotizing enterocolitis (NEC) | 120 Days of Life
Intracranial abnormalities | 120 Days of Life
Retinopathy of Prematurity (ROP) | 18-22 Months Corrected Age
Pulmonary hemorrhage | 120 Days of Life

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Schmidt, MD, Study Director — McMaster University; David K. Stevenson, MD, Principal Investigator — Stanford University; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University; Charles R. Bauer, MD, Principal Investigator — University of Miami; William Oh, MD, Principal Investigator — Brown University, Womens and Infants Hospital
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] Schmidt B, Davis P, Moddemann D, Ohlsson A, Roberts RS, Saigal S, Solimano A, Vincer M, Wright LL; Trial of Indomethacin Prophylaxis in Preterms Investigators. Long-term effects of indomethacin prophylaxis in extremely-low-birth-weight infants. N Engl J Med. 2001 Jun 28;344(26):1966-72. doi: 10.1056/NEJM200106283442602. PMID 11430325
- [Result] Schmidt B, Asztalos EV, Roberts RS, Robertson CM, Sauve RS, Whitfield MF; Trial of Indomethacin Prophylaxis in Preterms (TIPP) Investigators. Impact of bronchopulmonary dysplasia, brain injury, and severe retinopathy on the outcome of extremely low-birth-weight infants at 18 months: results from the trial of indomethacin prophylaxis in preterms. JAMA. 2003 Mar 5;289(9):1124-9. doi: 10.1001/jama.289.9.1124. PMID 12622582
- [Result] Ambalavanan N, Baibergenova A, Carlo WA, Saigal S, Schmidt B, Thorpe KE; Trial of Indomethacin Prophylaxis in Preterms (TIPP) Investigators. Early prediction of poor outcome in extremely low birth weight infants by classification tree analysis. J Pediatr. 2006 Apr;148(4):438-444. doi: 10.1016/j.jpeds.2005.11.042. PMID 16647401
- [Result] Schmidt B, Roberts RS, Fanaroff A, Davis P, Kirpalani HM, Nwaesei C, Vincer M; TIPP Investigators. Indomethacin prophylaxis, patent ductus arteriosus, and the risk of bronchopulmonary dysplasia: further analyses from the Trial of Indomethacin Prophylaxis in Preterms (TIPP). J Pediatr. 2006 Jun;148(6):730-734. doi: 10.1016/j.jpeds.2006.01.047. PMID 16769377
- [Result] Clyman RI, Saha S, Jobe A, Oh W. Indomethacin prophylaxis for preterm infants: the impact of 2 multicentered randomized controlled trials on clinical practice. J Pediatr. 2007 Jan;150(1):46-50.e2. doi: 10.1016/j.jpeds.2006.09.001. PMID 17188612
- [Result] Kabra NS, Schmidt B, Roberts RS, Doyle LW, Papile L, Fanaroff A; Trial of Indomethacin Prophylaxis in Preterms Investigators. Neurosensory impairment after surgical closure of patent ductus arteriosus in extremely low birth weight infants: results from the Trial of Indomethacin Prophylaxis in Preterms. J Pediatr. 2007 Mar;150(3):229-34, 234.e1. doi: 10.1016/j.jpeds.2006.11.039. PMID 17307535
- [Result] Alfaleh K, Smyth JA, Roberts RS, Solimano A, Asztalos EV, Schmidt B; Trial of Indomethacin Prophylaxis in Preterms Investigators. Prevention and 18-month outcomes of serious pulmonary hemorrhage in extremely low birth weight infants: results from the trial of indomethacin prophylaxis in preterms. Pediatrics. 2008 Feb;121(2):e233-8. doi: 10.1542/peds.2007-0028. PMID 18245398
- [Result] Bassler D, Stoll BJ, Schmidt B, Asztalos EV, Roberts RS, Robertson CM, Sauve RS; Trial of Indomethacin Prophylaxis in Preterms Investigators. Using a count of neonatal morbidities to predict poor outcome in extremely low birth weight infants: added role of neonatal infection. Pediatrics. 2009 Jan;123(1):313-8. doi: 10.1542/peds.2008-0377. PMID 19117897
- [Derived] Schmidt B, Seshia M, Shankaran S, Mildenhall L, Tyson J, Lui K, Fok T, Roberts R; Trial of Indomethacin Prophylaxis in Preterms Investigators. Effects of prophylactic indomethacin in extremely low-birth-weight infants with and without adequate exposure to antenatal corticosteroids. Arch Pediatr Adolesc Med. 2011 Jul;165(7):642-6. doi: 10.1001/archpediatrics.2011.95. PMID 21727276
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/